CLINICAL TRIAL: NCT01468675
Title: Health Information Technology (HIT) Enhanced Family History Documentation and Management in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jennifer S. Haas, MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009P002762
Record Dates: First submitted 2011-11-04; First posted 2011-11-09 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer; Breast Cancer; Coronary Heart Disease; Diabetes
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Coronary Disease; Diabetes Mellitus | interventions — Methods; Risk Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention is completion of a validated, web-based risk assessment used to assess personalized risk and generate a risk report
  Interventions: Other: Intervention
- Control (No Intervention): Usual Care

INTERVENTIONS:
Other: Intervention — risk assessment survey; decision support for providers for prevention based on risk
  Other Names: Risk Assessment and Prevention Recommendations
  Arms: Intervention

SUMMARY:
We evaluated whether collection of risk factors to generate an electronic health record (EHR)-linked personalized health risk appraisal (HRA) for coronary heart disease (CHD), diabetes, breast and colorectal cancer (CRC) was associated with improved patient-provider communication, risk assessment, and breast cancer screening plans in the next year.

DETAILED DESCRIPTION:
Growing evidence and understanding of an inherited component to several common, chronic diseases has led to an increase in the importance of information about family health history, and the integration of this information with other risk factors for common diseases, like lifestyle risk factors. The US Preventive Services Task Force (USPSTF) recommends the use of family health history as a routine genetic screening test for common diseases, as obtaining a complete family health history is the first step to identifying patients who are in need of intervention (e.g., intensive screening, lifestyle modification, preventative therapies, genetic counseling). The importance of integrating family health history with an individual's medical record will increase as our understanding of the genome evolves because it will be more essential to put detailed personal genetic information into a clinical context. Because of limited time during a typical primary care visit, and the concerns of primary care providers (PCPs) about their self-efficacy of estimating and providing guidance about risk, PCPs frequently do not obtain a family health history or provide individualized risk assessment. These issues highlight the need to leverage technology to collect these data independent of clinic visits, yet have these data interoperate with an individual's electronic health record (EHR). Telephonic interactive voice response systems (IVRS) and self-administered web-based tools are a low-cost, sustainable way of reaching out to primary care populations, independent of a visit. We propose to develop, implement, and evaluate a patient-reported, EHR-integrated personalized risk assessment module to provide tailored disease risk and risk reduction information.

The Specific Aims of the proposed project are to: Aim 1: Develop a patient-reported, EHR-integrated, personalized risk assessment module to provide tailored disease risk and risk reduction information for four common diseases (breast cancer, colorectal cancer, coronary heart disease, and type II diabetes) for the patient and his/ her PCP. Aim 2: Measure the reach and effectiveness of this integrated risk assessment module by conducting a cluster randomized controlled trial (RCT) of adult primary care patients in the Brigham and Women's Primary Care Practice-Based Research Network. Aim 3: Evaluate facilitators and barriers to the adoption and implementation of this integrated risk assessment module.

This project will further our understanding of how technology can be used to fill a gap in current clinical practice by facilitating the systematic collection of family health history and lifestyle risk factor data and integrating these data with an individual's EHR to personalize care in a variety of settings and for diverse patient populations. This work will use current national data standards for interoperability, and lessons learned from this project will be exportable to healthcare settings throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 - 75 Years old
* English or Spanish speaking
* Recent visit to a participating primary care practice

Exclusion Criteria

* No phone number or email address listed in the EHR

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6075 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Haas, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Risk Assessment and Prevention Recommendations
- Control: Control - Usual Care
Period: Overall Study
Arm/Group | Intervention | Control
Started | 2699 | 3376
Completed | 1699 | 2004
Not Completed | 1000 | 1372

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Risk Assessment and Prevention Recommendations provided to subjects
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 1699 | 2004 | 3703
Age, Continuous [Median (Full Range); unit: years] | 55 [18 to 75] | 56 [18 to 75] | 55 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1338 | 1415 | 2753
  Male | 361 | 589 | 950
Race/Ethnicity, Customized [Number; unit: participants]
  white | 1418 | 1675 | 3093
  black | 79 | 82 | 161
  Latino | 91 | 105 | 196
  Other/ unknown | 111 | 142 | 253
Region of Enrollment [Number; unit: participants]
  United States | 1699 | 2004 | 3703

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Discussed Disease Risk With Primary Care Provider
Time Frame: 3 months following primary care visit
Population: 1673+1847 (Total=3520) is the total number of subjects who answered the question that this outcome is derived from. (During your last doctor visit, did you talk to your PCP about your risk of developing cancer, heart disease or diabetes.) The total number of subjects included in the analysis is 3703.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Validated, web-based risk assessment is being used to assess personalized risk and generate a risk report
  risk assessment survey; decision support for providers for prevention based on risk
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1673 | 1847
Participants | 905 | 841

ADVERSE EVENTS:
Groups:
- Intervention: Intervention subjects completed a risk factors/perceptions assessment and received a 1 page Health Risk Assessment (HRA) prior to a primary care visit. This coded data was sent to the EHR. After their primary care visit, subjects again reported risk perception.
- Control: Control subjects completed a risk factors/perceptions assessment and received a 1 page Health Risk Assessment (HRA) AFTER their primary care visit. Coded data was not sent to the EHR.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/1699 | 0/2004
Serious Adverse Events (participants affected / at risk) | 0/1699 | 0/2004
Other Adverse Events (participants affected / at risk) | 0/1699 | 0/2004

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No